CLINICAL TRIAL: NCT04909346
Title: Observational Clinical Study of Anti-AAV Seroprevalence in Subjects With Ornithine Transcarbamylase Deficiency, Glycogen Storage Disorder Type Ia, and Wilson Disease
Brief Title: Adeno-Associated Virus (AAV) Antibody Study in Subjects OTC Deficiency, GSDIa, and Wilson Disease
Status: Terminated | Type: Observational
Why Stopped: Sponsor decision not related to safety concerns
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: UX431-CL001
Record Dates: First submitted 2021-05-26; First posted 2021-06-01 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Ornithine Transcarbamylase Deficiency; Wilson Disease; Glycogen Storage Disease Type IA
MeSH Terms: conditions — Ornithine Carbamoyltransferase Deficiency Disease; Hepatolenticular Degeneration; Hepatorenal form of glycogen storage disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and urine samples for future biomarker assay development
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this observational study is to evaluate the seroprevalence of anti-AAV antibodies in subjects with Ornithine Transcarbamylase (OTC) deficiency, Glycogen Storage Disease Type Ia (GSDIa), and Wilson Disease

DETAILED DESCRIPTION:
The study is primarily designed to follow a virtual model, in which Screening will take place over a telephone/video call. The study will comprise a single home health visit, either on the same day as Screening or within 30 days of enrollment. A safety follow-up may occur up to 5 days after Day 1 assessments are completed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of OTC deficiency, GSDIa, or Wilson Disease.
* Provide informed consent after the nature of the study has been explained, and prior to any research-related procedures.

Exclusion Criteria:

* Prior exposure to an AAV-based gene therapy.
* Concurrent or previous participation in another Ultragenyx clinical study.
* Recipient of a liver transplant.
* Presence or history of any condition that, in the view of the Investigator, would interfere with participation, pose undue risk, or would confound interpretation of results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will include approximately equal proportions of subjects with OTC deficiency, GSDIa, and Wilson Disease
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2021-06-23 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2022-11-17 (Actual)

PRIMARY OUTCOMES:
Prevalence of Anti-AAV8 Antibodies in Subjects with OTC Deficiency or GSDIa | Up to 35 days
Prevalence of Anti-AAV9 Antibodies in Subjects with Wilson Disease | Up to 35 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Ultragenyx Pharmaceutical Inc
Locations (5):
- Synexus Clinical Research US (Virtual Trial), Akron, Ohio, United States
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil
- McGill University Health Center, Montreal, Quebec, Canada
- Hospital Clínico Universitario de Santiago de Compostela, Santiago de Compostela, Spain
- Synexus North East Clinical Research Centre, Hexham, United Kingdom